CLINICAL TRIAL: NCT02488876
Title: Non-individual Related Ongoing Collection of Blood Samples for the Compilation of a Unique Database of Tissue Samples to Understand the Inflammatory Response After Cardiac Surgery
Brief Title: Database of Tissue Samples to Understand the Inflammatory Response After Cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: EK 151/09
Record Dates: First submitted 2015-05-04; First posted 2015-07-02 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Heart Diseases
Keywords: Cardiac surgery; Tissue sample database; Inflammatory responds
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to collect non-individual related blood samples for the compelling of a unique database of tissue samples to understand the inflammatory responds after cardiac surgery on an on-going basis. This includes especially protein analyses and genetic testing for certain neurotransmitters in the blood and tissues to understand disease markers related to heart disease. The study is designed as an openly recruiting biobank with the purpose to later serve multiple study purposes. Outcomes refer to protein analyses and genetic testing for neurotransmitters in the blood and tissues.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients scheduled for cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-04; Primary Completion 2099-12 (Estimated); Study Completion 2099-12 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Cytokines | Perioperatively until 7 days after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Goetzenich, PD Dr. med., Principal Investigator — Department of Cardiothoracic Surgery
Locations (1):
- University Hospital RWTH Aachen, Department of Thoracic and Cardiovascular Surgery, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Ney J, Heyland DK, Amrein K, Marx G, Grottke O, Choudrakis M, Autschbach T, Hill A, Meybohm P, Benstoem C, Goetzenich A, Fitzner C, Stoppe C. The relevance of 25-hydroxyvitamin D and 1,25-dihydroxyvitamin D concentration for postoperative infections and postoperative organ dysfunctions in cardiac surgery patients: The eVIDenCe study. Clin Nutr. 2019 Dec;38(6):2756-2762. doi: 10.1016/j.clnu.2018.11.033. Epub 2018 Dec 13. PMID 30583965